CLINICAL TRIAL: NCT07114796
Title: Nutritional Rehabilitation of Well Nourished Children With Persistent Diarrhea and Secondary Lactose Intolerance Using Rice Based Recipes Versus Already Prescribed Lactose Free Formulas .
Brief Title: Dietary Management of Well Nourished Children With Persistent Diarrhea and Secondary Lactose Intolerance With Different Feeding Formulas.( Hospital-Originated Modified Feeding HOMF)
Acronym: HOMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital and Institute of Child Health, Multan (Other Government)
Responsible Party: Principal Investigator, Dr. Saadia Khan, principal investigator, Children's Hospital and Institute of Child Health, Multan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1326-2819
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Ell-nourished Pediatric Patients; Nutritional Management in Diarrhea
Keywords: Persistent Diarrhea; Secondary Lactose Intolerance; Well-Nourished Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMMERCIAL LACTOSE FREE FORMULAS. (Active Comparator): feeding formula commercially available on 100 kcal per kg given ,1-1 dilution as per demand
  Interventions: Dietary Supplement: Standard Commercial Lactose-Free Formula
- Rice based recipe method feeding formula . (Experimental): rice based recipe method feed prepared at ward with rice oil,30 ml skimmed milk and sugar , given total of 100 kcal per kg of child on demand along rice based complementary feeding,
  Interventions: Dietary Supplement: Rice based recipe method feeding formula

INTERVENTIONS:
Dietary Supplement: Standard Commercial Lactose-Free Formula — "COMMERCIAL LACTOSE FREE FORMULAS" Intervention Type: Dietary Supplement or Nutritional Intervention
  Name of Intervention: Standard Commercial Lactose-Free Formula
  Description: A commercially available lactose-free formula (e.g., Isomil, Alfamino, or equivalent), used for feeding children during the stabilization phase of persistent diarrhea treatment.
  Route: Oral/Nasogastric
  Dosage: 130 ml/kg/day as per WHO schedule
  Duration: 7 days
  Arms: COMMERCIAL LACTOSE FREE FORMULAS.
Dietary Supplement: Rice based recipe method feeding formula — Rice based recipe method feeding formula" Intervention Type: Dietary Supplement or Nutritional Intervention
  Name of Intervention: Rice-Based Lactose-Free Therapeutic Formula
  Description: A locally prepared rice-based formula developed as an alternative to F-75, using puffed rice, sugar, oil, and micronutrient mix. It is lactose-free and used for feeding well-nourished children with persistent diarrhea.
  Route: Oral/Nasogastric
  Dosage: As per WHO feeding schedule - 130 ml/kg/day in 2-hourly feeds.
  Duration: 7 days during the stabilization phase
  For Arm: "COMMERCIAL LACTOSE FREE FORMULAS" Intervention Type: Dietary Supplement or Nutritional Intervention
  Name of Intervention: Standard Commercial Lactose-Free Formula
  Description: A commercially available lactose-free formula (e.g., Isomil, Alfamino, or equivalent), used for feeding children during the stabilization phase of persistent diarrhea treatment.
  Route: Oral/Nasogastric
  Dosage: 130 ml/kg/day as per WHO schedule
  Duration:
  Arms: Rice based recipe method feeding formula .

SUMMARY:
Interventional, treatment based study randomized control trial 32O Well nourished children allocated in 2 groups 160 each group ,Group A on lactose free commercial formula already in use,Group B ,ON Rice based feeding recipe .

DETAILED DESCRIPTION:
his clinical protocol is designed to evaluate and compare the effectiveness, safety, and acceptability of different feeding interventions in well-nourished pediatric patients diagnosed with persistent diarrhea (PD) complicated by secondary lactose intolerance (SLI). The study involves the administration of both commercial lactose-free formulas and hospital-originated, modified feeding recipes (HOMF), including rice-based porridge and protein-rich preparations, over a structured treatment duration.

Persistent diarrhea is defined as the passage of three or more abnormally loose or liquid stools per day, lasting more than 14 days, in the absence of other chronic gastrointestinal diseases. Secondary lactose intolerance is confirmed based on clinical presentation and stool findings such as acidic pH (<5.5) and positive reducing substances, typically resulting from post-infectious damage to the intestinal brush border where lactase activity resides.

The protocol consists of two parallel intervention arms:

Arm A (Formula-based group): Participants receive commercially available lactose-free pediatric formulas (LFFs) such as soy-based or hydrolyzed protein formulas, prepared as per manufacturer instructions. These formulas are age-appropriate, meet the caloric needs (~80-100 kcal/kg/day), and are devoid of lactose.

Arm B (Recipe-based group): Participants are administered locally-prepared therapeutic recipes standardized in the ward kitchen. Recipes include lactose-free rice milk, along with mung dal khichdi, and chicken broth-based porridges, designed for low osmolarity (<200 mOsm/L), high digestibility, and acceptable protein content. Recipes are prepared fresh daily under sterile conditions using pre-approved kitchen protocols and nutrient calculations.

All enrolled children are initially assessed for hydration status, weight, dietary history, and clinical signs of lactose intolerance. Baseline laboratory parameters (CBC, stool pH, reducing substances, electrolytes) are recorded. After informed consent, participants are randomized to either of the two intervention arms using block randomization (1:1 ratio), stratified by age and sex.

The feeding protocol is administered for 7-14 days, depending on clinical recovery and stool normalization. Feeding quantities are tailored based on caloric needs and tolerated volume, starting from 130 ml/kg/day and adjusted as per WHO guidelines for nutritional management in diarrhea. Monitoring includes daily stool frequency and consistency, weight changes, hydration status, adverse events, and acceptability of the diet (assessed by a 5-point hedonic scale).

Clinical improvement is defined as resolution of diarrhea (less than three loose stools per day), negative stool reducing substances, and normalization of stool pH (>6). If no improvement is observed by Day 5, re-evaluation is performed, and switching of the feeding strategy is considered only after safety clearance.

The study also explores the cost-effectiveness, caregiver acceptability, and preference patterns between the two approaches. Special attention is given to the preparation feasibility of the recipes in a home setting post-discharge, thereby promoting sustainability and local adaptability of therapeutic feeds in resource-limited environments.

All protocols follow ethical standards as per the Declaration of Helsinki and institutional IRB approval. The study is registered on a national trial registry. Data confidentiality is maintained using encrypted electronic records, and adverse events are reported in compliance with regulatory standards.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to hospital with persistent diarrhea and secondary lactose intolerance

Exclusion Criteria:

* less than 6months primary lactose intolerance critically ill children

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
stool frequency | day 1 to day 7 of feed
  episodes of loose stool per day

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad T Sultan, Phd, Study Chair — Bahuddin Zakariya University,Multan.
Locations (2):
- Pakistan (2):
  - Children's Hospital and Institute of child health Multan, Multan, Punjab Province
  - Tehsil Head Quater Sujah Abad, Multan Khurd, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This expert-consensus review (with clinical growth evidence) supports the use of hydrolyzed rice formulas as a first-line alternative to cow's milk-based eHF or AAF, showing adequate growth and high tolerability in infants (including well-nourished ones) — https://pubmed.ncbi.nlm.nih.gov/36438193/